CLINICAL TRIAL: NCT00239369
Title: A Prospective Randomised Study to Compare a Fixed Dose Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 25 mg With a Fixed Dose Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 12.5 mg in Patients With Uncontrolled Hypertension Who Fail to Respond Adequately to Treatment With a Fixed Dose Combination of Telmisartan 80 mg Plus Hydrochlorothiazide 12.5 mg
Brief Title: Telmisartan80/HCTZ25 Versus Telmisartan80/HCTZ12.5 in Hypertension Not Responding to Telmisartan80/HCTZ12.5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.480
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

INTERVENTIONS:
Drug: Fixed dose combination telmisartan 80 mg + HCTZ 25 mg
Drug: Fixed dose combination telmisartan 80 mg + HCTZ 12.5 mg

SUMMARY:
The primary objective of this trial is to demonstrate that a fixed dose combination of telmisartan 80 mg plus hydrochlorothiazide 25 mg (T80/H25) is superior in reducing blood pressure after eight weeks compared with a fixed dose combination of telmisartan 80 mg plus hydrochlorothiazide 12.5 mg (T80/H12.5) in patients who fail to respond to six weeks treatment with T80/H12.5.

DETAILED DESCRIPTION:
Adult patients with high blood pressure who are currently taking one, two or three blood pressure treatments will be asked to take part in the study. It is expected that about 1,600 patients in seventeen countries will enter the screening part of the study and approximately 480 of these patients will be allocated to double-blind randomised study treatment. The study will last for approximately fifteen weeks. Patients will visit the study doctor five times for assessment. After informed consent, patients will start a screening period for four to ten days. During the screening period, patients must take their usual blood pressure treatment but will stop this by the date of the next visit. If the patient is suitable for this study, they will then start run-in treatment period with telmisartan 80 mg plus hydrochlorothiazide 12.5 mg (T80/H12.5) taken as a single tablet once per day for approximately six weeks.

At the end of the run-in treatment period, if the diastolic blood pressure (DBP) is below 90 mmHg, the patient will not proceed as their blood pressure is already controlled by T80/H12.5. If the DBP is 90 mmHg or greater they will start the randomised study treatment period and be randomly allocated to double-blind treatment with either telmisartan 80 mg plus hydrochlorothiazide 25 mg(T80/H25) or T80/H12.5 taken as a single tablet once per day for eight weeks. They will also receive a placebo tablet (a dummy tablet which contains no active ingredient) every day.

They will visit the clinic four weeks and eight weeks later for assessment of their blood pressure and general health. Their participation in the study is complete eight weeks after the start of the randomised treatment period.

Study Hypothesis:

The trial hypothesis is that the reduction in seated trough DBP (i.e., seated trough DBP at the end of the randomised treatment period compared with the seated trough DBP at the start of the randomised treatment period) will be greater in the T80/H25 group compared with the T80/H12.5 group.

Comparison(s):

The efficacy and safety of the two trial treatments (T80/H25 versus T80/H12.5) will be compared. Trough blood pressure is the blood pressure 24 hours after the last dose of trial medication.

ELIGIBILITY:
Inclusion criteria:

* Essential hypertension.
* Currently taking between one and three antihypertensive medications at a stable dose for at least four weeks before Visit 1.
* Blood pressure not adequately controlled on existing treatment before entry (inadequate control defined as seated DBP >= 95 mmHg on one current antihypertensive medication or DBP >= 90 mmHg on two or more current antihypertensive medication(s).
* Failure to respond to six weeks treatment with T80/H12.5. (Failure to respond defined as seated DBP >= 90 mmHg at six weeks. This criterion will be assessed at Visit 3.)
* Willing and able to provide written informed consent.

Exclusion criteria:

* Women of child-bearing potential NOT practising acceptable means of birth control, positive serum pregnancy test, breastfeeding.
* Known or suspected secondary hypertension.
* Mean SBP >= 200 mmHg.
* Severe hepatic or renal impairment.
* Bilateral renal artery stenosis (or in a solitary kidney), post-renal transplant or only one functioning kidney.
* Clinically relevant hypokalaemia or hyperkalaemia.
* Uncorrected volume or sodium depletion, primary aldosteronism.
* Hereditary fructose intolerance.
* Previous symptoms of angioedema after ACE inhibitors or angiotensin-II receptor antagonists.
* Drug or alcohol dependency within the previous six months.
* Administration of any medication known to affect blood pressure.
* Concurrent participation in another clinical trial or any investigational therapy.
* Hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve.
* Allergic hypersensitivity to any component of the formulations under investigation.
* Concomitant therapy with lithium, cholestyramine or colestipol resins. non-compliance with study medication (less than 80% or more than 120%) during th e run-in treatment period.
* Any other clinical condition which, in the opinion of the investigator, would not allow safe administration of telmisartan or hydrochlorothiazide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08

PRIMARY OUTCOMES:
Change from baseline in trough seated DBP | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in trough seated SBP | 8 weeks
Change from baseline in trough standing DBP and SBP | 8 weeks
The proportion of patients achieving DBP control (trough seated DBP<90 mmHg). | 8 weeks
The proportion of patients achieving DBP response (trough seated DBP<90 mmHg or trough seated DBP reduction from baseline ≥10 mmHg). | 8 weeks
The proportion of patients achieving SBP response (trough seated SBP<140 mmHg or trough seated SBP reduction from baseline ≥10 mmHg). | 8 weeks
The proportion of patients achieving SBP response (trough seated SBP<140 mmHg or trough seated SBP reduction from baseline ≥20 mmHg) | 8 weeks
The proportion of patients in trough seated BP categories: opt.: SBP<120 mmHg and DBP<80 mmHg., norm.: SBP<130 mmHg and DBP<85 mmHg and not optimal, high-normal: SBP<140 mmHg and DBP<90 mmHg and not optimal or normal, high: SBP ≥140 mmHg or DBP ≥90 mmHg | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BIL UK / Ireland
Locations (74):
- Denmark (5):
  - Boehringer Ingelheim Investigational Site, Birker?d
  - Boehringer Ingelheim Investigational Site, Haderslev
  - Boehringer Ingelheim Investigational Site, Odder
  - Boehringer Ingelheim Investigational Site, R?dovre
  - Boehringer Ingelheim Investigational Site, Vildbjerg
- Finland (4):
  - Boehringer Ingelheim Investigational Site, Helsinki
  - Boehringer Ingelheim Investigational Site, Joensuu
  - Boehringer Ingelheim Investigational Site, Kokkola
  - Boehringer Ingelheim Investigational Site, Turku
- France (3):
  - ALTI, Angers
  - Hopital Avicenne, Bobigny
  - Mg Recherches, Paris
- Germany (8):
  - Boehringer Ingelheim Investigational Site, Ellefeld
  - Boehringer Ingelheim Investigational Site, Flörsheim
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Ingelheim
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
- Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- Ireland (8):
  - Boehringer Ingelheim Investigational Site, Birr
  - Boehringer Ingelheim Investigational Site, Carrigallen
  - Boehringer Ingelheim Investigational Site, Dublin
  - Boehringer Ingelheim Investigational Site, Enniscorthy
  - Boehringer Ingelheim Investigational Site, Gorey
  - Boehringer Ingelheim Investigational Site, Mallow
  - Boehringer Ingelheim Investigational Site, New Ross
  - Boehringer Ingelheim Investigational Site, Toomyvara
- Italy (4):
  - Ospedale Arnaboldi, Broni (PV)
  - Azienda Ospedaliera Universita di Ferrara, Ferrara
  - IRCCS San Raffaele, Roma
  - Ospedale Civile, Vittorio Veneto (TV)
- Boehringer Ingelheim Investigational Site, Kuching, Sarawak, Malaysia
- Netherlands (9):
  - Boehringer Ingelheim Investigational Site, Bennebroek
  - Boehringer Ingelheim Investigational Site, Ewijk
  - Boehringer Ingelheim Investigational Site, Helmond
  - Boehringer Ingelheim Investigational Site, Hoogwoud
  - Boehringer Ingelheim Investigational Site, Nijverdal
  - Boehringer Ingelheim Investigational Site, Oude Pekela
  - Boehringer Ingelheim Investigational Site, Rijswijk
  - Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - Boehringer Ingelheim Investigational Site, Rotterdam
- Norway (5):
  - Boehringer Ingelheim Investigational Site, Elverum
  - Boehringer Ingelheim Investigational Site, Moelv
  - Boehringer Ingelheim Investigational Site, Oslo
  - Boehringer Ingelheim Investigational Site, Skedsmokorset
  - Boehringer Ingelheim Investigational Site, Tolvsr?d
- South Africa (7):
  - Boehringer Ingelheim Investigational Site, Bellville
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Lenasia
  - Boehringer Ingelheim Investigational Site, Lenasia South
  - Boehringer Ingelheim Investigational Site, Midrand
  - Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (2):
  - Boehringer Ingelheim Investigational Site, Incheon
  - Boehringer Ingelheim Investigational Site, Seoul
- Spain (8):
  - Hospital Municipal de Badalona, Badalona / Barcelona
  - Hospital de Galdakao, Galdakao / Vizcaya
  - Hospital Gral. Jerez de la Frontera, Jerez de La Frontera / Cadiz
  - C.A.P. Mosen Cinto Verdaguer, L'Hospitalet de Llobregat / Barcelona
  - Hospital Universitario Gregorio Mara?on, Madrid
  - C.A.P. Ronda Cerdanya, Mataro (Barcelona)
  - Hospital General de Mostoles - Medicina Interna, Mostoles / Madrid
  - Hospital del Conxo, Santiago de Compostela
- Sweden (4):
  - Boehringer Ingelheim Investigational Site, Eksjö
  - Boehringer Ingelheim Investigational Site, Karlstad
  - Boehringer Ingelheim Investigational Site, Uddevalla
  - Boehringer Ingelheim Investigational Site, Uppsala
- Switzerland (4):
  - Boehringer Ingelheim Investigational Site, Basel
  - Boehringer Ingelheim Investigational Site, Bellinzona
  - Boehringer Ingelheim Investigational Site, Saint-Imier
  - Boehringer Ingelheim Investigational Site, Vezia
- Boehringer Ingelheim Investigational Site, Taipei, Taiwan

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/18772643